CLINICAL TRIAL: NCT00128791
Title: Intracoronary Nitroprusside for the Prevention of the No-Reflow Phenomenon Following Primary Percutaneous Coronary Intervention in Acute Myocardial Infarction. A Randomized, Double Blind, Placebo-Controlled Clinical Trial
Brief Title: Nitroprusside for Prevention of no-Reflow in Primary Angioplasty
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: sor323102ctil
Record Dates: First submitted 2005-08-09; First posted 2005-08-10 (Estimated); Last update posted 2007-05-25 (Estimated); Status verified 2007-05

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; angioplasty; nitric oxide; prevention; acute myocardial infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Nitroprusside

INTERVENTIONS:
Drug: Nitroprusside

SUMMARY:
In patients admitted with acute myocardial infarction, there is a total occlusion of a coronary artery. Even after emergency catheterization and angioplasty, in some patients, the resumed blood flow is suboptimal and impacts on heart function. The study is aimed at examining whether nitroprusside, an anti-hypertension medication, given directly into the coronary artery, can improve the blood flow after the removal of the obstruction that caused the infarction.

DETAILED DESCRIPTION:
Inadequate myocardial tissue perfusion despite successful relief of the culprit occlusion and restoration of epicardial coronary flow for ST-segment elevation acute myocardial infarction (STEMI) results in poor outcome. The investigators hypothesized that nitroprusside (NTP) injected intracoronary immediately before angioplasty might prevent no-reflow and improve vessel flow and myocardial perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Acute ST elevation myocardial infarction (MI) patients planned for primary PCI
* Diagnostic angiography demonstrating a TIMI flow grade <3 in the coronary artery before the PCI

Exclusion Criteria:

* An admission electrocardiogram (ECG) showing complete left bundle branch block or a paced rhythm
* Systolic blood pressure < 90 mmHg
* A history of coronary bypass operation
* A known allergic reaction to nitroprusside
* Chronic hemodialysis
* Intravenous drug abuse
* Pregnancy
* Rescue intervention after failed thrombolysis
* Contraindications to aspirin or clopidogrel
* Need for emergent coronary artery bypass surgery
* Inability to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2003-01; Study Completion 2005-04

PRIMARY OUTCOMES:
The coronary blood flow in the artery undergoing intervention following angioplasty as determined by the corrected Thrombolysis in Myocardial Infarction (TIMI) frame count (CTFC)
Proportion of patients with complete ST-segment resolution immediately after percutaneous coronary intervention (PCI)

SECONDARY OUTCOMES:
The proportion of patients with TIMI grade 3 flow after the procedure
The proportion of patients with myocardial grade 3 blush after the procedure
The proportion of patients with complete ST-segment resolution at 24 hours post intervention
The proportion of patients requiring intra-aortic balloon counter-pulsation and its duration of use
Length of hospital stay
The combined rate of target vessel revascularization, myocardial infarction or death at 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Doron Zahger, MD, Principal Investigator — Soroka UMC, Beer-sheva, Israel
Locations (1):
- Soroka University Medical Center, Beersheba, Israel